CLINICAL TRIAL: NCT06580457
Title: Understanding and Treating Substance Use Disorder and Comorbid Conditions in Veterans' Real-Life Settings
Brief Title: Personalized Approach to Healthy Use and Recovery (PATH) Trial
Acronym: PATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Emory University (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURA-009-24S; 1IK2CX002716 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder
Keywords: substance use disorder; precision medicine; ecological momentary assessment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Receive the personal causal model with a 1-hour, live clinical feedback session.
  Interventions: Behavioral: Personal Causal Model + Personalized Feedback
- Control (No Intervention): No clinical feedback session. Personal causal models will be provided at the end of the study for those who wish to receive them.

INTERVENTIONS:
Behavioral: Personal Causal Model + Personalized Feedback — Receive a personal causal model of one's personalized causes of substance use/urges, along with a 1-hour, live clinical feedback session to suggest how to apply these insights to one's own recovery.
  Arms: Intervention

SUMMARY:
An important part of substance use treatment for many people is learning what triggers their substance use and urges, and how they can better manage those triggers. In this study, the investigators will generate a model for each individual that shows likely causal links between their substance use, urges, and comorbid symptoms (e.g., anxiety, depression, and PTSD), and the investigators will examine these models as a group to draw conclusions about common causes for substance use (and recovery) among Veterans with substance use disorders. The investigators will also test whether receiving a personal model and clinical feedback improves substance use disorder and comorbid symptom outcomes. Results will include both patient-reported and statistically-determined causes of substance use for individuals and groups, clinical impact of a personalized model and feedback session, and participant feedback about the relevance of this study and intervention.

DETAILED DESCRIPTION:
Substance use disorders (SUDs) are very common in Veterans, with 1 in 3 Veterans meeting criteria for a SUD each year. SUDs typically occur in the context of other comorbid conditions, such as depressive disorders, post-traumatic stress disorder (PTSD), or anxiety disorders. For Veterans who have comorbid conditions and SUD, treatment outcomes are worse than those who have SUD only. The investigators propose that the factors leading to poor SUD treatment outcomes in this population are not adequately understood and, based on preliminary research, vary widely by individual. The investigators propose to measure SUD and comorbid symptoms multiple times daily in Veterans with SUD to characterize the connections between SUD and comorbid conditions for each individual. N = 74 Veterans with SUD will complete personalized 4-week ecological momentary assessment (EMA) protocols measuring SUD and comorbid symptoms, as well as personalized items relevant to each Veteran's presentation. Personalized models will be estimated from each Veteran's EMA data using causal discovery analyses. Veterans will be randomized to either intervention or control groups. The intervention group will receive their personal causal models along with an hour-long clinical feedback session based on their model. The investigators will also attempt to integrate the models into any ongoing treatment and deliver follow-up reminders of key insights from their models to the intervention participants throughout the remainder of the study. Follow-up measures will assess the impact of receiving this personalized intervention. A subset of N = 24 Veterans who were in the intervention group will be invited to share their feedback on the acceptability, relevance, and usefulness of the EMA protocol, personal models, and clinical feedback, as well as thoughts on the factors that support recovery versus problematic substance use. Specific aims are: 1) to identify the momentary causes of substance use and urges for Veterans with SUD, both individually and as a group, 2) Examine the clinical impact of receiving personal causal models of substance use and urges, and 3) Refine the personal causal models and clinical feedback to improve acceptability and relevance to Veterans. This project will advance understanding of day-to-day maintenance mechanisms for problematic substance use in Veterans with SUD. This study will create causal models of substance and comorbid symptoms at the individual level and test the impact of receiving clinical feedback based on these models. Aims will be accomplished through a training plan that involves conducting VA clinical trials, using causal discovery, and using qualitative analyses to leverage feedback from participants.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study are intended to include most Veterans with SUD
* inclusion criteria are current probable SUD as indicated by:

  * a clinical score on the alcohol use disorders identification test (AUDIT) or drug use disorders identification test (DUDIT)
  * past-month substance use
  * a reliable access to a smartphone, tablet, or other device with capability of accessing and completing surveys throughout the day

    * this will exclude those who are currently completing inpatient treatment

Exclusion Criteria:

* exclusion criteria are being under the influence of a judgment-impairing substance at the time of consent (e.g., cannabis, alcohol, illicit opioids)

  * participants will be invited to return another day
* being legally compelled to complete treatment
* or being under civil commitment

  * due to lack of ability to give autonomous consent in these situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
Substance use | 4-, 8-, and 12-week follow-ups
  Substance use will be measured as number of days each substance was used in the past 30 days using National Survey on Drug Use and Health questions. Substances measured are nicotine, alcohol, cannabis, cocaine/crack, heroin, hallucinogens, inhalants, methamphetamine, pain relievers, tranquilizers, sedatives, and prescription stimulants. For alcohol, we will also obtain number of drinks consumed on each day, and will analyze whether average number of drinks per drinking day has changed during each follow-up period.
Substance-related problems | 4-, 8-, and 12-week follow-ups
  Substance-related problems will be measured for the past month using the Alcohol Use Disorders Identification Test (AUDIT) and Drug Use Disorders Identification Test (DUDIT). Scores range from 0 to 40. Scores will be analyzed for changes at each follow-up point.

SECONDARY OUTCOMES:
PTSD Symptoms | 4-, 8-, and 12-week follow-ups
  PTSD Checklist 5 or PCL-5 measures past 30 day PTSD symptoms. Scores range from 0 to 80. Scores will be analyzed for changes at each follow-up point.
Anxiety Symptoms | 4-, 8-, and 12-week follow-ups
  Generalized Anxiety Disorder (GAD-7) measures anxiety symptoms over the last 2 weeks. Scores range from 0 to 21. Scores will be analyzed for changes at each follow-up point.
Depression Symptoms | 4-, 8-, and 12-week follow-ups
  Beck Depression Inventory (BDI) measures depression symptoms over the last month. Scores range from 0 to 63. Scores will be analyzed for changes at each follow-up point.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Stevenson, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
A deidentified, anonymized dataset will be created and shared.